CLINICAL TRIAL: NCT05872308
Title: Hemorrhagic Myocardial Infarction Detection With High-sensitivity Cardiac Troponin-I
Brief Title: Hemorrhagic Myocardial Infarction Detection by Post-reperfusion Troponin Kinetics
Acronym: MIRON-TROP
Status: Completed | Type: Observational
Sponsor: Rohan Dharmakumar (Other)
Responsible Party: Sponsor-Investigator, Rohan Dharmakumar, Vice Chair of Research, Medical Imaging Research Institute, Indiana University School of Medicine
Organization: Indiana University (Other)
Other Study IDs: 13081
Record Dates: First submitted 2023-05-14; First posted 2023-05-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Acute Myocardial Infarction
Keywords: STEMI; Troponin; Intramyocardial Hemorrhage; Cardiac MRI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pilot trial to determine diagnostic efficacy of post-reperfusion troponin kinetics in detection of hemorrhagic myocardial infarction

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Index STEMI
3. Coronary angiogram with PCI to occur irrespective of the onset of the symptoms.
4. Ability to provide informed consent for themselves

Exclusion Criteria:

1. History of prior myocardial infarction,
2. Cardiogenic shock,
3. Patients who present with current cardiac arrest
4. Any contraindication to cardiac CMR (claustrophobia, pacemaker or cardiac defibrillator, known allergy to gadolinium),
5. Presence of permanent atrial fibrillation,
6. Unconscious patient,
7. Severe renal insufficiency (creatinine clearance ≤ 30 ml/min/m2 or renal replacement therapy),
8. Women who are pregnant or breastfeeding. Women of reproductive potential must have a negative pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals aged 18 to 80 who have been diagnosed with acute ST-elevation myocardial infarction (STEMI) and are scheduled for emergency percutaneous coronary intervention (PCI).
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Diagnostic Threshold | 48 hours
  Levels of markers in hemorrhagic infarct vs. non-hemorrhagic infarct

SECONDARY OUTCOMES:
Peak levels of serum troponin-I | 48 hours
  peak levels of serum troponin-I in hemorrhagic infarct vs non-hemorrhagic infarct
Area under the curve (AUC) for serum troponin-I | 48 hours
  area under the curve post-MI for troponin-I
Hemorrhagic infarct size | 48 hours
  as determined by cardiac MRI
Hemorrhagic infarct volume | 48 hours
  as determined by cardiac MRI
Hemorrhagic infarct microvascular obstruction | 48 hours
  as determined by cardiac MRI
Hemorrhagic infarct area at risk | 48 hours
  as determined by cardiac MRI

CONTACTS AND LOCATIONS:
Overall Officials: Keyur P Vora, MD FACC, Principal Investigator — Faculty
Locations (2):
- IU Methodist Hospital, Indianapolis, Indiana, United States
- Synergy Cardiovascular Research Center, Synergy Superspecialty Hospital, Rajkot, Gujarat, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vora KP, Kalra A, Shah CD, Bhatt K, Kumar A, Pandya T, Poptani V, Chan SF, Singh D, Jambunathan N, Subramanian R, Youssef K, Kanakasabai S, Finney R, Desai A, Kreutz RP, Kovacs RJ, Raman SV, Bhatt DL, Dharmakumar R. In-Hospital Mortality in Hemorrhagic Myocardial Infarction. NEJM Evid. 2025 Sep;4(9):EVIDoa2400294. doi: 10.1056/EVIDoa2400294. Epub 2025 Aug 26. PMID 40858097